CLINICAL TRIAL: NCT05947981
Title: Is Pre-operative Infusion of 5% Dextrose Effective in Reducing the Incidence of PONV in Middle Ear Surgery? A Blinded Randomized Control Trial
Brief Title: Pre-operative 5% Dextrose Infusion & PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shymaa Fathy, Assistant professor of anesthesia and SICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MS-206-2022
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Nausea, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Glucose; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Patients will be fasted and not receiving any pre-operative fluids
- Dextrose group (Active Comparator): Patients will take 100ml/HR of clear fluids (apple juice) during the fasting hours till 2 hrs before the operation and will receive dextrose 5% infusion at a rate of 1ml/kg/h 2hrs before the operation and till the end of the operation
  Interventions: Dietary Supplement: Dextrose 5%, normal saline
- Normal saline group (Placebo Comparator): Patients will take 100ml/HR of water during the fasting hours till 2 hrs before the operation and will receive normal saline 0.9% at a rate of 1ml/kg/h (group NS) intravenously (IV)2hrs before the operation and till the end of the operation
  Interventions: Dietary Supplement: Dextrose 5%, normal saline

INTERVENTIONS:
Dietary Supplement: Dextrose 5%, normal saline — Decrease fasting hours
  Arms: Dextrose group; Normal saline group

SUMMARY:
With this study, we aim to compare the efficacy of pre-operative dextrose-containing fluid infusion with other fluid for the prevention of PONV in middle ear surgeries.

DETAILED DESCRIPTION:
We hypothesized that maintenance of stable level of blood glucose in addition to adequate hydration through preoperative intravenous dextrose 5% infusion will have a rule in decreasing the incidence and severity of PONV; as it reduces insulin resistance and decreases gastric acid secretion; which may contribute to PONV.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and ll.
* Patients undergoing middle ear surgeries, mastoidectomy, or tympanoplasty

Exclusion Criteria:

* history of dependence or use of antiemetics
* history of motion sickness
* presence of psychiatric illness
* pregnant and lactating women
* cardiovascular disorders (Ischemic heart diseases, congestive heart failure and valvular diseases)
* Diabetic patients

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
PONV | 24 hours
  incidence

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine- Cairo University, Cairo, Egypt